CLINICAL TRIAL: NCT06387290
Title: Optimizing Chronic Pain Care With Mindfulness and Chronic Pain Management Visits
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Principal Investigator, Eric Garland, Professor, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00172836
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Prescription Opioid Misuse; Substance-Related Disorders; Pain; Narcotic-Related Disorders; Chemically-Induced Disorders; Mental Disorders; Opioid-Related Disorders; Neurologic Manifestations
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Substance-Related Disorders; Pain; Narcotic-Related Disorders; Chemically-Induced Disorders; Mental Disorders; Neurologic Manifestations

STUDY DESIGN:
Intervention Model Description: Hybrid implementation-effectiveness trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators, study staff, and statistician will be blinded to treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Oriented Recovery Enhancement + Patient-centered chronic pain management visits (Experimental): Participants will attend a Mindfulness-Oriented Recovery Enhancement (MORE) group weekly for eight weeks, in addition to patient-centered chronic pain management visits led by their primary care provider.
  Interventions: Behavioral: Mindfulness Oriented Recovery Enhancement; Behavioral: Patient-Centered Chronic Pain Management Visits
- Patient-centered chronic pain management visits (Active Comparator): Participants will attend patient-centered chronic pain management visits led by their primary care provider.
  Interventions: Behavioral: Patient-Centered Chronic Pain Management Visits

INTERVENTIONS:
Behavioral: Mindfulness Oriented Recovery Enhancement — Mindfulness-Oriented Recovery Enhancement (MORE) is a group behavioral intervention that unites mindfulness training, cognitive reappraisal, and positive psychological principles into an integrative therapeutic approach.
  Arms: Mindfulness Oriented Recovery Enhancement + Patient-centered chronic pain management visits
Behavioral: Patient-Centered Chronic Pain Management Visits — Participant will meet with their primary care provider for patient-centered care and shared decision making while discussing their chronic pain management strategy (e.g., opioid analgesics).

SUMMARY:
The primary aim of this implementation-effectiveness trial is to examine the effectiveness of Mindfulness-Oriented Recovery Enhancement (MORE) and patient-centered chronic pain management visits in primary care as interventions to reduce chronic pain, improve quality of life, and reduce opioid-related harms among chronic pain patients on long-term opioid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 +
* Current chronic pain diagnosis (pain for ≥3 months) determined by physician assessment
* Prescribed long-term opioid therapy (≥3 months)
* Score >=3 on the Pain Enjoyment General Activity scale
* Score >=9 on the Current Opioid Misuse Measure OR lifetime psychiatric or substance use disorder diagnosis OR benzodiazepine use OR history of overdose OR patient or physician determination that risks of opioid use may outweigh the benefits of opioid use

Exclusion Criteria:

* Chronic pain due to a cancer diagnosis
* Active suicidal intent, schizophrenia, psychotic disorder
* Prior experience with Mindfulness-Based Stress Reduction, Mindfulness-Based Cognitive Therapy, Mindfulness-Based Relapse Prevention, or Mindfulness-Oriented Recovery Enhancement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Misuse | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Opioid misuse as evidenced by triangulated aggregate of self-reported Current Opioid Misuse Measure and/or interview via Addiction Behaviors Checklist and/or urine screen
Chronic Pain | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Change in Chronic pain will be measured from baseline through study completion using the Pain, Enjoyment of Life, and General Activity Scale (PEG). Scoring can be determined in one of two ways:
  1. A total sum score from 0 to 30, with higher scores indicating more severe pain and pain-related interference with life and activities
  2. Dividing the sum of responses to all three items by 3 to get the mean score on a scale of 0-10, with higher scores indicating more severe pain and pain-related interference with life and activities.

SECONDARY OUTCOMES:
Change in Quality of Life | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Change in Quality of Life will be measured from baseline through study completion using the Patient Reported Outcomes Measurement Information System (PROMIS-29) to assess physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity. Scores range from 4-20 in each domain, with higher scores indicating more impairment in that domain.
Opioid Dosing | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Opioid dose will be assessed from baseline through study completion by Timeline Follow Back (TLFB) interview. Opioid dose will be converted to morphine-equivalent using equianalgesic conversions.
Opioid Craving | Daily from baseline through month 4
  Opioid craving will be assessed with validated numeric rating scale items (Garland et. al, 2022) delivered by ecological momentary assessment.
PTSD Symptoms | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  PTSD Symptoms will be measured from baseline through study completion using the Posttraumatic Stress Disorder Checklist (PCL-5). Scores range from 0-80, with higher scores indicating overall higher PTSD symptom severity.
Depression | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Depression symptoms will be measured from baseline through study completion using the nine-item Patient Health Questionnaire (PHQ-9). Scores range from 0-27, with higher scores indicating more severe symptoms of depression.
Generalized Anxiety | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Generalized Anxiety will be measured from baseline through study completion using the Generalized Anxiety Disorder 7 (GAD-7). Scores range from 0-21, with higher scores indicating more severe symptoms of anxiety.

OTHER OUTCOMES:
Decentering | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Change in Decentering from baseline through study completion will be measured with the Metacognitive Processes of Decentering (MPODS) scale. Scores range from 15 to 75, with higher scores indicating more decentering.
Mindful Reappraisal of Pain Sensations | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Change in Mindful Reappraisal of Pain Sensations from baseline through study completion will be assessed with the Mindful Reappraisal of Pain Sensations (MRPS) Scale. Scores range from 0 to 54, with higher scores indicating greater mindful reappraisal of pain sensations.
Savoring | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Change in savoring measured by the Brief Savoring Inventory, range from 4 to 20, higher scores indicating more use of savoring.
Reappraisal | Change from baseline through study completion (assessed at 3-, 6-, 9-, and 12-months follow-up)
  Change in reappraisal measured by the Emotion Regulation Questionnaire, range from 6 to 42, with a higher score indicating more use of reappraisal.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCSD Health, La Jolla, California
  - Rutgers University Primary Care Clinics, New Brunswick, New Jersey
  - University of Utah Primary Care Clinics, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will conform to National Institutes of Health (NIH) regulations and our resource sharing plan
Supporting Information: Study Protocol, ICF
Time Frame: At the time with publication of the primary outcome results